CLINICAL TRIAL: NCT03302702
Title: A Comparison Trial of Eight Weeks Versus Twelve Weeks of Exercise Program in Interstitial Lung Diseases.
Brief Title: Duration of Exercise Program in Interstitial Lung Diseases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof, Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKC4
Record Dates: First submitted 2017-10-01; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Interstitial Lung Disease
Keywords: exercise; duration
MeSH Terms: conditions — Lung Diseases, Interstitial; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise program (Other): Treatment group
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — Exercise program including breathing control, pursed-lip breathing, diaphragmatic and thoracic breathing, aerobic and strengthening training

SUMMARY:
We aimed to compare the functional results of the 8th week with the results of the 12th week of the exercise programs applied to the patients with ILD.

DETAILED DESCRIPTION:
Exercise programs (EP) have been shown to be the effective approach for functional outcomes in interstitial lung diseases (ILD). In many studies, the duration of exercise programs varies between 8-12 weeks. However, the optimal duration of exercise program is still unknown.

We aimed to compare the results of the 8th week with the results of the 12th week of the PR programs applied to the patients with ILD.

A total of 14 patients with ILD referred to our PR unit [11 idiopathic pulmonary fibrosis, 2 sarcoidosis (stage 3 and 4) and 1 nonspecific interstitial pneumonia] were included in the study. Pulmonary function test, arterial blood gas analysis, 6- minute walk test, mMRC dyspnea scale, quality of life questionnaires and hospital anxiety depression scale were performed before, at the 8th and 12th weeks after the exercise program applied to the patients twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 12 week exercise program
* Diagnosed with ILD

Exclusion Criteria:

* Not completed 12 week exercise program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | 6 minute
  It was performed in a 30-meter long corridor in accordance with American Thoracic Society criteria

SECONDARY OUTCOMES:
mMRC | 5 minutes
  It was used for dyspnea that patients felt during their daily activities.
Pulmonary Function Test | 20 minutes
  It was used for assessment of lung functions
SGRQ | 30 minutes
  A disease-specific quality of life scale
SF-36 Health Survey | 30 minutes
  A health related quality of life scale
Hospital Anxiety and Depression Inventory | 20 minutes
  It was used for assessment of anxiety and depression

IPD SHARING:
Plan to Share IPD: No